CLINICAL TRIAL: NCT00885222
Title: Antidepressant Effect of Deep Brain Stimulation (DBS) in Parkinson's Disease (PD) Patients: Relationship of Stimulation Parameters to Improvement in the Clinical Features of Depression in PD Patients.
Brief Title: Antidepressant Effect of Deep Brain Stimulation in Parkinson's Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr Renana Eitan, MD., Hadassah Medical Organization, Jerusalem, Israel
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Eitan-DBS-PD-MDD-HMO-CTIL
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-05

CONDITIONS: Parkinson's Disease; Major Depressive Disorder
Keywords: Parkinson's disease; Major depressive disorder; Deep brain stimulation
MeSH Terms: conditions — Parkinson Disease; Depressive Disorder, Major

ARMS (3):
- 1 (Active Comparator): PD patient that were treated with STN DBS and developed depression after the surgery (n=5).
  Interventions: Device: DBS parameters setting
- 2 (Active Comparator): PD patients with depression that are candidates for STN DBS (n=5).
  Interventions: Device: DBS parameters setting
- 3 (Active Comparator): PD patients without depression that are candidates for STN DBS (n=10).
  Interventions: Device: DBS parameters setting

INTERVENTIONS:
Device: DBS parameters setting — DBS parameters will be set to increase the DBS affected volume to include both the cognitive and limbic territories in addition to the dorso-lateral motor territories of the STN. This novel approach to parameter selection is directed to achieve improvement in cognitive and limbic as well as motor domains of PD. The patients will therefore be assessed for cognitive, limbic and motor state at multiple time points; there will be a baseline assessment prior to starting treatment (prior to DBS surgery and/or prior to parameters changes); thereafter assessments will follow the stimulation parameter changes; thereafter follow-up assessments at 6 - 12 months. Stimulation parameters will be changed every 2 weeks or earlier if an urgent clinical state emerges. Patients with depression will be monitored for antidepressant effects of stimulation changes. Patients without depression will be monitored for evidence of treatment emergent depression.

SUMMARY:
The purpose of this study is:

1. To determine, in the context of a prospective clinical trial, whether stimulation parameters in PD patients treated with DBS, are associated with antidepressant effects.
2. To determine whether these antidepressant effects are related to or independent of changes in the motor features of PD.
3. To establish a computerized database that includes stimulation parameters and clinical parameters in PD patients treated with DBS.
4. To develop a computer-assisted decision making protocol for programming of DBS parameters in both depressed and non-depressed PD patients.

DETAILED DESCRIPTION:
Depressive symptoms of PD patients are major predictors of their prognosis and quality of life. Therefore, successful treatment of depression is crucial in PD patients. Using deep brain stimulation as an antidepressant (or to augment a standard antidepressant) could be a promising new direction. The hypothesis to be tested in the current project is that treatment with deep brain stimulation will improve both the neurological and the psychiatric (depressive) symptoms of PD. It is further hypothesized that the improvement in depressive symptoms will not be a simple consequence of improvement in neurological status. Data from this open label study will form the basis for planning a larger scale controlled trial in depressed PD patients and exploratory studies in patients with major depression who do not have PD.

Today, programming of DBS is based on the neurological evaluation of the motor features of PD. If our hypothesis is proven, i.e. parameter manipulation of DBS affects the mental features of PD, it is crucial to establish a valid database that will enable to study these effects. Moreover, such a detailed database will be the basis for the development of a computer-assisted decision making protocol for programming of DBS. A novel decision making protocol will maximize the benefits of DBS in both depressed and non-depressed PD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically definite PD treated / candidates for treatment with DBS (patients with advanced idiopathic PD who are deemed appropriate for DBS surgery).
2. Patients will be included in the study irrespective of whether a diagnosis of major depression (mild to moderate but not severe MDD) is fulfilled at baseline. Patients without depression will be monitored in the study for evidence of treatment emergent depression. Patients with depression will be monitored for antidepressant effects of stimulation change.
3. Age 40-75 years
4. Male or female.
5. Competent and willing to give written informed consent.

Exclusion Criteria:

1. Significant suicidal risk [Hamilton Depression scale item 3 (suicide) >2].
2. Comorbidity with any Psychotic Disorder, Bipolar Disorder, Post Traumatic Stress Disorder (PTSD), Eating Disorder.
3. Lifetime history of substance or alcohol dependence or of abuse in the preceding 12 months
4. Significant cognitive decline, as measured by Addenbrooke's Cognitive Examination (ACE) and the Frontal Assessment Battery (FAB).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure of the study will be the stimulation parameters of patients who fulfill criteria for MDD at the inception of trial and manifest remission (HAM-D21 score <7) after 4 months (or less) of DBS treatment. | 18 months

SECONDARY OUTCOMES:
Secondary outcome measures will be the relationship between improvement in mental status (as measured by HAM-21, BDI, CGI, HAM-A, BPRS and PDQ39) and change in PD symptoms (as measured by UPDRS). | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Renana Eitan, MD, Principal Investigator — Hadassah Medical Organization; Zvi Israel, MD, Study Chair — Hadassah Medical Organization; Hagai Bergman, MD, Study Chair — Hadassah Medical Organization; Bernard Lerer, MD, Study Chair — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel